CLINICAL TRIAL: NCT06540014
Title: The Difference of Weight Gain Tendencies During Pregnancy According to Pregestational Body Mass Indices of the Mothers in Two Different Ethnic Populations- Does it Make Difference Regarding Neonatal Outcomes?
Brief Title: The Difference of Weight Gain Tendencies and Obesity During Pregnancy
Status: Completed | Type: Observational
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Suzan Sahin, associate professor, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: BucaSeyfiDemirsoyRTH
Record Dates: First submitted 2024-07-27; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Obesity, Maternal; Weight Gain, Maternal; Birth Weight; Birth Outcome, Adverse
Keywords: Maternal obesity; neonatal outcome; weight gain in pregnancy; immigrant; Syrian; Turkish
MeSH Terms: conditions — Pregnancy in Obesity; Gestational Weight Gain; Birth Weight; Pregnancy Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Turkish: Belonging to Turkish race originally
  Interventions: Other: No intervention
- Syrian: Belonging to Syrian race originally
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is made, groups are formed just due to the races.

SUMMARY:
Background: Excess weight and obesity are a global pandemic, particularly among women of childbearing age. Pre-pregnancy obesity is linked to adverse maternal and neonatal outcomes, including preterm birth, macrosomia, stillbirth, and neonatal death. These risks vary by maternal age, race, and ethnicity, with rising rates among immigrant and minority women. This study investigates overweight and obesity rates in pregnant women, weight gain during pregnancy, and adherence to guidelines and possible neonatal outcomes, comparing Turkish and Syrian immigrant women.

Methods: This retrospective single-center study was conducted at Buca Seyfi Demirsoy Teaching and Research Hospital in Izmir, Turkey, over one year. Data collected included demographic information, pregnancy complications, delivery modes, maternal and neonatal anthropometric measurements, and neonatal morbidity and mortality. The study included Turkish and Syrian women with complete medical records. Statistical analyses were performed using SPSS software, with significance set at p < 0.05.

DETAILED DESCRIPTION:
Background: Excess weight and obesity are a global pandemic, particularly among women of childbearing age. Pre-pregnancy obesity is linked to adverse maternal and neonatal outcomes, including preterm birth, macrosomia, stillbirth, and neonatal death. These risks vary by maternal age, race, and ethnicity, with rising rates among immigrant and minority women. This study investigates overweight and obesity rates in pregnant women, weight gain during pregnancy, and adherence to guidelines and possible neonatal outcomes, comparing Turkish and Syrian immigrant women.

Methods: This retrospective single-center study was conducted at Buca Seyfi Demirsoy Teaching and Research Hospital in Izmir, Turkey, over one year. Data collected included demographic information, pregnancy complications, delivery modes, maternal and neonatal anthropometric measurements, and neonatal morbidity and mortality. The study included Turkish and Syrian women with complete medical records. Statistical analyses were performed using SPSS software, with significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Being admitted to our hospital for delivery or having just given birth
* Being Turkish or Syrian
* Having all detailed information, including mothers' pregestational and immediate pre-delivery body weights, available in medical records

Exclusion Criteria:

* Significant deficiencies in medical records
* Belonging to an ethnic group other than Turkish or Syrian

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In the study, the hospital records of all pregnant women admitted for delivery at the obstetrics ward of the Women's and Children's Diseases additional service building Buca Seyfi Demirsoy Training and Research Hospital were retrospectively reviewed over a 6-month period from September 1, 2022, to February 28, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Maternal weight gain | 1 year period until inclusion
  Total body weight gained by pregnant women during pregnancy according to the measurements made by "Tanita" scale

SECONDARY OUTCOMES:
Obesity and overweight | 6 months
  Pregestational obesity or being overweight

OTHER OUTCOMES:
Neonatal morbidities | 6 months
  Neonatal morbidities experienced by the babies
Adherence to the weight gain guidelines | 6 months
  Adherence to the recommendations of current guidelines regarding total body weight gain according to the measurements made by "Tanita" scale

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Şahin, Assoc.Prof., Study Director — Izmir Democracy University
Locations (1):
- Buca Seyfi Demirsoy RTH, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hung TH, Hsieh TT. Pregestational body mass index, gestational weight gain, and risks for adverse pregnancy outcomes among Taiwanese women: A retrospective cohort study. Taiwan J Obstet Gynecol. 2016 Aug;55(4):575-81. doi: 10.1016/j.tjog.2016.06.016. PMID 27590385
- [Result] Zhao R, Xu L, Wu ML, Huang SH, Cao XJ. Maternal pre-pregnancy body mass index, gestational weight gain influence birth weight. Women Birth. 2018 Feb;31(1):e20-e25. doi: 10.1016/j.wombi.2017.06.003. Epub 2017 Jul 14. PMID 28716548
- [Result] Heslehurst N, Ells LJ, Simpson H, Batterham A, Wilkinson J, Summerbell CD. Trends in maternal obesity incidence rates, demographic predictors, and health inequalities in 36,821 women over a 15-year period. BJOG. 2007 Feb;114(2):187-94. doi: 10.1111/j.1471-0528.2006.01180.x. PMID 17305899